CLINICAL TRIAL: NCT01239719
Title: Randomized Study for Effectiveness and Safety Evaluation of Dexamethasone 0.5 mg + Fumarate Clemastine 1 mg Compared to Dexamethasone 0.5 mg in Patients With Allergic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clínica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DECEMS11209; Version 02 - Amendment 02
Record Dates: First submitted 2010-04-08; First posted 2010-11-11 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Allergy; Dermatitis
Keywords: Allergic dermatitis
MeSH Terms: conditions — Hypersensitivity; Dermatitis; Dermatitis, Atopic | interventions — clemastine, dexamethasone drug combination; Dexamethasone

ARMS (2):
- Dexamethasone + Clemastine (Experimental): Dexamethasone + clemastine fumarate cream
  Interventions: Drug: Dexamethasone + clemastine
- Dexamethasone (Active Comparator): Dexamethasone 0.5 mg
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone + clemastine — Dexamethasone 0.5 mg clemastine fumarate: 01 tablet every 12 hours.
  Arms: Dexamethasone + Clemastine
Drug: Dexamethasone — Dexamethasone 0.5 mg: 01 tablet every 12 hours.
  Arms: Dexamethasone

SUMMARY:
The aim of this study is to prove the efficacy of the dexamethasone 0.5 mg + 1 mg clemastine fumarate tablet compared to 0.5 mg of dexamethasone in reducing the signs and symptoms of allergic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the IC in two ways, agreeing with all study procedures
* Patients aged above 18 years of any ethnicity, class or social group, female or male
* Patients with acute, subacute or chronic dermatoses, of inflammatory and / or allergic origin, to which it is recommended the use of drugs under investigation, such as:

  * atopic dermatitis
  * prurigo
  * primary contact dermatitis or allergic hives
  * drug eruption
  * allergic vasculitis
  * dyshidrosis, Note: The above clinical conditions are diagnosed from clinical examination.

Exclusion Criteria:

* Patients being treated with antibiotics
* Participation in clinical trials in the 12 months preceding the investigation
* Current treatment with immunosuppressants (eg, cyclosporine or methotrexate)
* Current treatment with phototherapy (UVA, UVB, PUVA and lasers)
* Use of systemic corticosteroids in the visit to include or 15 days preceding the survey
* Topical treatments at the site of lesions in the 15 days preceding the survey
* Presence of any skin condition
* Presence of secondary infections at the site of treatment, diagnosed clinically;
* Presence of other eczematous diseases, such as nummular eczema, neurodermatitis, seborrheic dermatitis, psoriasis, scabies, and Buckley's syndrome
* Pregnant or lactating women
* Chronic alcoholism
* Patients with a history of hypersensitivity to any component of the products under investigation.
* Any finding of clinical observation (clinical history or physical examination) that is interpreted by the physician investigator as a risk to the patient's participation in the study.
* Allergic Dermatosis mild or, acording to the investigator criteria, is not justified systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate, through clinical examinations, the effectiveness of the combination tablet with 0.5 mg of dexamethasone and clemastine 1 mg, compared with 0.5 mg tablet of dexamethasone in improving the signs and symptoms associated with allergic dermatitis. | 14 days of treatment.
  Evaluating the effectiveness of the polypill dexamethasone 0.5 mg + 1 mg clemastine fumarate tablet compared to 0.5 mg of dexamethasone in improvement of signs (erythema, edema and lesion length) and symptoms (itching) associated with frames of dermatoses allergic.

SECONDARY OUTCOMES:
Evaluation of the efficacy. | 14 days of treatment.
  Constitute secondary signals of efficacy including excoriation, oozing, crusting and lichenification.